CLINICAL TRIAL: NCT00337454
Title: A Phase I/II Study of BMS-354825 in Subjects With Imatinib Resistant or Intolerant Philadelphia Chromosome Positive Chronic Myelogenous Leukemia and Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia Who Are Resistant or Intolerant to Treatment
Brief Title: Study of BMS-354825 in Subjects With CML Who Are Resistant to or Intolerant of Imatinib or Ph+All in Japan
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA180-031
Record Dates: First submitted 2006-06-14; First posted 2006-06-16 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: Imatinib resistant or intolerant CML; Treatment resistant or intolerant Ph+ALL
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Dasatinib

ARMS (6):
- A1 (Experimental)
  Interventions: Drug: Dasatinib
- A2 (Experimental)
  Interventions: Drug: Dasatinib
- A3 (Experimental)
  Interventions: Drug: Dasatinib
- B1 (Experimental)
  Interventions: Drug: Dasatinib
- B2 (Experimental)
  Interventions: Drug: Dasatinib
- B3 (Experimental)
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Tablets, Oral, 50mg BID, once daily, 24 weeks.
  Other Names: Sprycel
  Arms: A1
Drug: Dasatinib — Tablets, Oral, 70mg BID, once daily, 24 weeks.
  Other Names: Sprycel
  Arms: A2
Drug: Dasatinib — Tablets, Oral, 90mg BID, once daily, 24 weeks.
  Other Names: Sprycel
  Arms: A3
Drug: Dasatinib — Tablets, Oral, 70mg BID, once daily, 24 weeks.
  Other Names: Sprycel
  Arms: B1
Drug: Dasatinib — Tablets, Oral, 70mg BID, once daily, 12 weeks.
  Other Names: Sprycel
  Arms: B2
Drug: Dasatinib — Tablets, Oral, 70mg BID, once daily, 12 weeks.
  Other Names: Sprycel
  Arms: B3

SUMMARY:
This study is composed of Phase I and Phase II part. Phase I part: The objective is to evaluate the safety of BMS-354825 in subject with chronic phase Chronic Myelogenous Leukemia (CML). Dosage of BMS-354825 will be 50 mg BID, 70 mg BID or 90 mg BID. Phase II part: The objective is to evaluate the efficacy of BMS-354825. dosage will be decided according to the results of Phase I part. Treatment period will be 6 months for subjects with chronic phase CML, and 3 months for subjects with accelerated phase or blast phase CML and Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia (Ph+ALL)

ELIGIBILITY:
Inclusion Criteria:

* Philadelphia chromosome positive or bcr-abl gene positive
* Chronic Myelogenous Leukemia (CML)
* Subjects must have primary or acquired resistance to imatinib mesylate or have intolerance of imatinib mesylate
* Philadelphia Chromosome Positive Acute Lymphoblastic leukemia (Ph+ALL)
* Subjects must have primary or acquired resistance to chemotherapy or have intolerance of chemotherapy
* Performance status (general conditions) specified by the Eastern Cooperative Oncology Group: 0-2
* Men and women, ages 20 - 75
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 3 months after the study in such a manner that the risk of pregnancy is minimized

Exclusion Criteria:

* Subjects who are eligible and willing to undergo transplantation at pre-study
* Women who are pregnant or breastfeeding
* Uncontrolled or significant cardiovascular disease
* History of significant bleeding disorder unrelated to CML or ALL
* Adequate hepatic function
* Adequate renal function
* Medication that increase bleeding risk
* Medication that change heart rhythms
* Subjects who are compulsorily detained for legal reasons or treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study

Ages: 20 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2005-07; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of BMS-354825 administered orally twice daily for 4 weeks, evaluate the efficacy of BMS-354825 as defined by cytogenetic response for subjects with chronic phase CML, and as defined by hematologic response

SECONDARY OUTCOMES:
Pharmacokinetic profiles, cytogenetic response and hematologic response, BCR-ABL point mutations and biochemical assays of BCR-ABL, safety, time to and duration of hematologic and cytogenetic response
response

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (18):
- Japan (18):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Maebashi, Gunma
  - Local Institution, Nishinomiya-Shi, Hyōgo
  - Local Institution, Kagoshima, Kagoshima-ken
  - Local Institution, Isehara-Shi, Kanagawa
  - Local Institution, Kanagawa, Kanagawa
  - Local Institution, Kyoto, Kyoto
  - Local Institution, Sendai, Miyagi
  - Local Institution, Nagasaki, Nagasaki
  - Local Institution, Okayama, Okayama-ken
  - Local Institution, Moriguchi, Osaka
  - Local Institution, Iruma-Gun, Saitama
  - Local Institution, Hamamatsu, Shizuoka
  - Local Institution, Tochigi, Tochigi
  - Local Institution, Bunkyo-Ku, Tokyo
  - Local Institution, Chuo-Ku, Tokyo
  - Local Institution, Shinjuku-Ku, Tokyo
  - Local Institution, Tokyo, Tokyo